CLINICAL TRIAL: NCT02077621
Title: The Phase II Clinical Study of PG2 Injection for Improving Fatigue in Patients After Palliative Abdominal Surgery for Cancer
Brief Title: Study of PG2 Injection for Improving Fatigue in Patients After Palliative Abdominal Surgery for Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study reevaluation
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PH-CP020
Record Dates: First submitted 2014-02-24; First posted 2014-03-04 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Surgery; Fatigue
Keywords: cancer-related fatigue; Palliative Abdominal Surgery; HRQL
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PG2 (Experimental): Treatment Group:
  PG2 (500 mg in 500 ml saline), 1 dose a day before surgery and 1 dose a day for 3 days after surgery
  Interventions: Drug: PG2
- Placebo (Placebo Comparator): Control group:
  Placebo (500 ml saline), 1 dose a day before surgery and 1 dose a day for 3 days after surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PG2 — Powder for Injection, 500 mg PG2/500 ml normal saline
  Other Names: PG2 injection 500mg
  Arms: PG2
Drug: Placebo — 500 mL normal saline
  Arms: Placebo

SUMMARY:
PG2 has been approved in Taiwan to treat cancer-related fatigue for advanced cancer patients. The primary objective of this study is to evaluate the efficacy of PG2 on fatigue relief in patients undergoing palliative abdominal surgery for cancer. The secondary endpoints, including the length of hospital stay, postoperative complications, HRQL, inflammatory biomarkers, the duration of antibiotic therapy, mortality during the hospital stay, weight loss and body composition, will be evaluated among these patients.

DETAILED DESCRIPTION:
This will be a double-blind, randomized, and placebo-controlled study. At least 40 evaluable patients who are scheduled for palliative abdominal surgery for cancer will be randomly assigned to the control or treatment group. Each group will have at least 20 patients and be treated as follows: 1) control group: patients will accept placebo 1 dose a day (POD-1) before surgery and 1 dose a day for 3 days after surgery (POD+0 to POD+2); 2) treatment group: patients will accept PG2 1 dose a day (POD-1) before surgery and 1 dose a day for 3 days after surgery (POD+0 to POD+2).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have cancer and are scheduled for palliative abdominal surgery for cancer
* Age > 20 years older
* Patients who signed the informed consent form

Exclusion Criteria:

* Patients, at screening, has levels greater than 2.5 times the upper limit of normal liver function of alanine aminotransferase or aspartate aminotransferase.
* Patients has a severe renal impairment (defined as serum creatinine greater than 2 times the upper limit of normal or BUN greater than 2.5 times the upper limit of normal for range); or the subject is on dialysis.
* Patients have ongoing infection, respiratory tract dysfunction, cardiac dysfunction or immune disorder that, in the opinion of the investigator, may interfere with conduct of the study.
* Patients who are not suitable for undergoing surgery (e.g. congenital hemostatic disorders) by the investigator's judgment.
* Patients have enrolled or have not yet completed other investigational drug trials within 1 month before screening.
* Female patients are pregnant or breast-feeding.
* Patients who require preoperative nutritional support
* Patients with serious comorbidities (American Society of Anesthesiologists Risk Class of 4 or 5).
* Patients who is unwilling or unable to answer the quality of life questionnaires i.e. the BFI-T and EORTC QLQ-C30.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
change from baseline fatigue status | a day before surgery and day 1,2,7,28,56,84 after surgery
  qustionnaires

SECONDARY OUTCOMES:
Length of hospital stay | 13 weeks
Postoperative complications | 13 weeks
  patients were observed for surgical and nonsurgical complication
Health-related Quality of Life (HRQL) | a day before surgery and for day 7,28,56,84 after surgery
Inflammatory biomarkers: Serum IFN-r, IL-1b, IL-4, IL-6, IL-10 and TNF-a | Before operation and on day 1, and day 7 after operation
The duration of antibiotic therapy | 13 weeks
Mortality during the hospital stay | 13 weeks
Weight loss | 13 weeks
  patients will be measured during follow-up period
Body composition | a day before surgery and for day 28 after surgery
  such as protein, mineral, body fat mass

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ming Wu, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided